CLINICAL TRIAL: NCT06499285
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Elritercept (KER-050) for the Treatment of Transfusion-Dependent Anemia in Adult Participants With Very Low-, Low-, or Intermediate-Risk Myelodysplastic Syndromes (MDS) (RENEW)
Brief Title: A Study of Elritercept to Treat Anemia in Adults With Very Low, Low, or Intermediate Risk Myelodysplastic Syndromes (MDS) Who Need Regular Blood Transfusions
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KER-050-D301; 2024-516009-22-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Myelodysplastic Syndromes
Keywords: Anemia; Elritercept; Myelodysplastic neoplasms; KER-050; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 2:1 ratio to receive either elritercept (TAK-226, KER-050) or placebo, respectively, subcutaneously every 4 weeks. Randomization will be stratified according to ring sideroblast status and baseline transfusion burden.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study in which treatment assignment will be blinded for the Participant, care provider, Investigators and any personnel (other than the selected unblinded personnel) involved with the study conduct or evaluation at the investigational sites, the CRO, and the Sponsor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elritercept (Experimental): Participants will be administered elritercept (TAK-226, KER-050), subcutaneously every 4 weeks, up to 48 weeks or until the end of treatment period.
  Interventions: Drug: Elritercept
- Placebo (Placebo Comparator): Participants will be administered elritercept (TAK-226, KER-050) matching-placebo, subcutaneously every 4 weeks, up to 48 weeks or until the end of treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Elritercept — Elritercept (TAK-226, KER-050) administered subcutaneously every 4 weeks.
  Other Names: KER-050; TAK-226
  Arms: Elritercept
Drug: Placebo — Elritercept (TAK-226, KER-050) matching-placebo administered subcutaneously every 4 weeks.
  Arms: Placebo

SUMMARY:
The main aim of this study is to find out how well elritercept works in lowering the need for RBC transfusions. Other aims are to learn how well elritercept works in reducing the need for RBC transfusions over longer periods of time or in adults with high transfusion needs. The study will also check on how safe elritercept is and how well it is tolerated.

DETAILED DESCRIPTION:
This is a Phase 3, double-blind, randomized, placebo-controlled study to evaluate the efficacy and safety of elritercept (TAK-226, KER-050) versus placebo. Elritercept (TAK-226, KER-050) is an investigational medicinal product being developed for the treatment of anemia in adult participants with a diagnosis of lower-risk myelodysplastic neoplasms/syndromes. After all required Screening Period assessments are completed, and eligibility is confirmed, participants will be randomized and enter the Primary Phase of the Double-Blind Treatment Period. Participants will be randomly assigned in a 2:1 ratio to receive either elritercept (TAK-226, KER-050) or placebo subcutaneously (SC) every 4 weeks (Q4W). Participants will be stratified according to their RS status (RS-positive versus non-RS) and baseline transfusion burden (LTB versus HTB). The Primary Phase of the Double-blind Treatment Period will last 24 weeks. The Secondary Phase of the Double-Blind Treatment Period will last an additional 24 weeks. During the Secondary Phase of the Double-Blind Treatment Period, all participants will continue to receive the same double-blind treatment they received during the Primary Phase. Study visits will occur approximately every 2 weeks from Cycle 1 through Cycle 6 and every 4 weeks from Cycle 7 through the remainder of the Double-Blind Treatment Period. During the Extension Phase of the Double-Blind Treatment Period, all eligible participants will continue to receive the same double-blind treatment they received during the Primary and Secondary Phases. Participants will continue in the Extension Phase until they individually discontinue or until the study is unblinded. For participants to remain on double-blind treatment, they must meet the criteria outlined in the MDS disease assessment criteria every 24 weeks. Based on the outcome of the Week 24 MDS disease assessment, participants will either continue in the Extension Phase of the Double-blind Treatment Period or will be discontinued from treatment and proceed to End of Treatment and then into the Safety Follow-up Period. The Safety Follow-Up Period will extend from the last dose of study treatment through 8 weeks after the last dose of study treatment. Study visits should occur every 4 weeks within the Safety Follow-Up Period. Long-term follow-up will take place quarterly after a participant has completed the Safety Follow-Up Period. Long-term follow-up will continue for 5 years from the first dose of study treatment or 3 years after the last dose, whichever is longer, or until a participant is deceased, is lost to follow-up, withdraws consent, or the study closes, whichever is earliest.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information and/or protected personal data in accordance with national and local study participant data protections and privacy regulations.
* Male or female greater than or equal to (≥)18 years of age at the time of signing informed consent.
* Diagnosis of MDS with or without RS (as determined in an evaluable bone marrow aspirate, read by an independent central reader to confirm diagnosis at Screening) according to the World Health Organization 2016 classification that meets the International Prognostic Scoring System-Revised (IPSS-R) classification of very low, low, or intermediate risk disease.
* Transfusion dependence assessed in the 16 weeks immediately preceding randomization in two 8-week blocks, classified as either:

  a. Low-transfusion burden (LTB), defined as 4 to 7 red blood cells (RBC) units per 16 weeks; or b. High-transfusion burden (HTB), defined as ≥8 RBC units per 16 weeks; and c. For all participants: i. Only transfusion events for a pretransfusion hemoglobin (Hgb) lesser than (<)10 grams per deciliter (g/dL) are counted toward eligibility; ii. At least 1 transfusion event in each 8-week period and a minimum of 2 transfusion events separated by ≥7 days within the 16-week period immediately preceding randomization; and iii. No consecutive 56-day period can be RBC transfusion-free during the 16-week period immediately preceding randomization.
* Refractory or intolerant to prior erythropoiesis-stimulating agent (ESA) treatment (discontinued ≥4 weeks before randomization), or unlikely to respond to ESA treatment, defined as follows:

  a. Refractory to prior ESA treatment: documentation of nonresponse or a response that was no longer maintained with a prior ESA-containing regimen, either as a single agent or combination (e.g., with granulocyte colony-stimulating factor [G-CSF]); ESA regimen must have been either: i. Recombinant human erythropoietin (EPO) ≥40,000 international units per week (IU/week) for ≥8 doses or equivalent; or ii. Darbepoetin alpha ≥500 micrograms (μg) every 3 weeks for ≥4 doses or equivalent.

  b. Intolerant to prior ESA treatment: documentation of discontinuation of a prior ESA-containing regimen, either as a single agent or combination (e.g., with G-CSF), at any time after introduction due to intolerance or an AE.

  c. Unlikely to respond to ESA treatment: low chance of response to ESA based on an endogenous serum EPO level greater than (>)200 units per liter (U/L).
* Less than 5% blasts in an evaluable bone marrow aspirate collected at Screening, read by an independent central reader.
* Eastern Cooperative Oncology Group performance status of 0 to 2.
* Females of childbearing potential and sexually active males must agree to use highly effective methods of contraception.
* In the opinion of the Investigator, the participant is able and willing to comply with the requirements of the protocol (e.g., all study procedures, return for follow-up visits).

Exclusion Criteria:

* Del(5q) MDS or therapy-related (secondary) MDS.
* Anemia due to any other known cause (e.g., thalassemia, hemolytic anemia, bleeding events, or deficiency of iron, B12, and/or folate).
* Receipt of RBC transfusion for any reason(s) other than underlying MDS within 16 weeks before randomization.
* Clinically significant cardiovascular disease defined as:

  1. New York Heart Association heart disease class III or IV;
  2. Fridericia corrected QT (QTcF) interval >500 milliseconds during Screening;
  3. Presence of uncontrolled hypertension defined as mean systolic blood pressure ≥160 millimeters of mercury (mm Hg) or diastolic blood pressure ≥100 mm Hg during Screening; or
  4. Uncontrolled arrhythmia, myocardial infarction, or unstable angina within 6 months before Screening.
* Known ejection fraction <35%, confirmed by a local echocardiogram performed during Screening, or a previously performed echocardiogram if collected within 6 months before Screening.
* Child-Pugh class C hepatic impairment.
* Stroke, deep vein thrombosis, or pulmonary embolism within 6 months before Screening.
* Any known history of acute myeloid leukemia (AML).
* Prior history of malignancies, other than MDS, unless participant has been free of the disease (including completion of any treatment, including maintenance, for prior malignancy) for ≥ 5 years. However, participants with a history or concurrent diagnosis of the following conditions are allowed if not requiring systemic therapy:

  1. Basal or squamous cell carcinoma of the skin;
  2. Carcinoma in situ of the cervix;
  3. Carcinoma in situ of the breast; and/or
  4. Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, node, metastasis [TNM] clinical staging system).
* History of solid organ or bone marrow transplantation.
* Active infection requiring intravenous treatment (e.g., antibiotics, antifungals, or antivirals) within 28 days, or oral treatment within 14 days before randomization.
* History of or known active chronic infection with HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV). Participants without known positive history of HIV, HBV, and/or HCV do not require further testing, unless testing is mandated per local guidelines.
* Body mass index ≥ 40 kilograms per meter square (kg/m^2).
* Major surgery within 28 days before randomization.
* History of allergy/anaphylaxis to investigational medicinal product (IMP) excipients (refer to the current elritercept IB for a list of excipients) or recombinant proteins.
* Prior use of elritercept, luspatercept, or sotatercept.
* Prior use of hypomethylating agents (HMAs), isocitrate dehydrogenase inhibitor, lenalidomide, imetelstat, or immunosuppressive therapy given for treatment of MDS.
* Iron chelation therapy initiated within 8 weeks before randomization. Participants on stable doses of iron chelation therapy for ≥ 8 weeks are allowed.
* Vitamin B12 or folate therapy initiated within 4 weeks before randomization. Participants on stable replacement doses for ≥ 4 weeks and without ongoing concurrent vitamin B12 or folate deficiency are allowed.
* Androgen use within 8 weeks before randomization. Participants on stable androgen dosing for hypogonadism for ≥ 8 weeks are allowed.
* High-dose corticosteroid use within 4 weeks before randomization. Participants on stable chronic steroid doses of prednisone lesser than or equal to (≤) 10 mg/day or corticosteroid equivalent for ≥ 4 weeks are allowed.10 mg/day or corticosteroid equivalent for ≥ 4 weeks are allowed.
* Treatment with any investigational drug within 28 days before Screening or, if the half-life of the product is known, within 5 times the half-life before Screening, whichever is longer.
* Ongoing participation in another interventional clinical study.
* Serum EPO level >500 U/L.
* Platelet count ≥450 × 10^9/L or ≤25 × 10^9/L.
* Absolute neutrophil count ≤ 500/µL.
* Serum aspartate aminotransferase or alanine aminotransferase ≥3 × the upper limit of normal (ULN).
* Total bilirubin ≥2 × ULN unless attributable to Gilbert's syndrome.
* Ferritin ≤ 50 micrograms per litre (μg/L).
* Folate ≤2.0 nanograms per milliliter (ng/mL).
* Vitamin B12 ≤200 picograms per milliliter (pg/mL).
* Estimated glomerular filtration rate <30 milliliters per minute per 1.73 meter square (mL/min/1.73m^2) as determined by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Collaboration equation.
* Pregnant or lactating female.
* Any other condition not specifically noted above that, in the opinion of the Investigator, would preclude the participant from participating in the study or could confound interpretation of data from the study.
* Investigational site staff members directly involved in the conduct of the study and site staff members otherwise supervised by the Investigator, employees of the Sponsor or contract research organization (CRO) directly involved in the conduct of the study, or immediate family members (defined as a spouse, parent, child, or sibling, whether biological or legally adopted).
* For Participants in France: Persons under court protection, persons not affiliated with a social security system, and protected adults (per applicable French law [Art. L. 1121-6, Art. L. 1121-8, Art. L. 1121-8-1]).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2032-05-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Transfusion Independence (TI) for ≥8 Weeks | Baseline through Week 24
  Transfusion independence is defined as the absence of any red blood cells (RBC) transfusions in a period of at least 8 weeks after the first dose of the study treatment through week 24.

SECONDARY OUTCOMES:
Percentage of Participants Achieving TI for ≥24 Weeks | Baseline through Week 48
  Transfusion independence is defined as the absence of any RBC transfusions in a period of at least 24 weeks after the first dose of the study treatment through week 48.
Percentage of Participants with High-transfusion Burden (HTB) Achieving TI for ≥8 weeks | Baseline through Week 24
  Transfusion independence is defined as the absence of any RBC transfusions in a period of at least 8 weeks after the first dose of the study treatment through week 24.
Number of Participants with Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From the time of signing the informed consent form through 60 days after the last dose of study treatment, approximately 6 years
  An adverse event (AE) is defined as any untoward medical occurrence, in a clinical study participant administered a medicinal product, that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not it is related to study treatment. A TEAE is defined as an AE that commences on or after the first dose of the study treatment and within 60 days after the last dose of the study treatment, or analysis cutoff date, whichever is earlier. An SAE is any untoward medical occurrence that, at any dose: results in death, is life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a medically important event.
Change from Baseline in Clinical Laboratory Values, Vital Signs, and Electrocardiograms (ECGs) | From the time of signing the informed consent form through safety follow-up, approximately 16 months
  Change from baseline in clinical laboratory values, vital signs, and ECGs will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (156):
- United States (21):
  - City of Hope, Duarte, California
  - Los Angeles Cancer Network, Glendale, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - University of Miami Hospital and Clinics, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - ILCC. Illinois Cancer Centers, Peoria, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Maryland Oncology Hematolofy, Columbia, Maryland
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Clinical Research Alliance NY, Westbury, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - Cleveland Clinic - Cleveland, Cleveland, Ohio
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Baptist Clinical Research Institute, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology Northeast Texas, Denison, Texas
  - U.T. MD Anderson Cancer Center, Division of Cancer Medicine, Houston, Texas
  - Texas Oncology Gulf Coast, The Woodlands, Texas
  - Tranquil Research, Webster, Texas
- Australia (7):
  - Westmead Hospital, Sydney, New South Wales
  - Townsville University Hospital, Douglas, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - St Vincent's Hospital (Melbourne) Ltd, Fitzroy, Victoria
  - Peter MacCallum Cancer Center, Parkville, Victoria
- Brazil (8):
  - Porto Alegre Clinical Hospital (HCPA), Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus, Clinical Research Unit - Cancer Institute, Porto Alegre, Rio Grande do Sul
  - Pontifical University Of Rio Grande Do Sul (PUCRS) - St. Luke Hospital, Porto Alegre, Rio Grande do Sul
  - Sao Jose do Rio Preto Regional Faculty of Medicine Foundation, São José do Rio Preto, São Paulo
  - Americas Institute, Rio de Janeiro
  - Portuguese Charity of Sao Paulo, Clinical Hematology / Oncology Center, São Paulo
  - Hospital A.C.Camargo ("Antonio Prudente" Foundation), São Paulo
  - Santa Casa of Mercy of Santos, São Paulo
- Bulgaria (5):
  - Dr. Pencho Georgiev - Outpatient Center for Individual Practice for Specialized Medical Care in Internal Medicine and Clinical Hematology (EOOD), Plovdiv
  - University Multiprofile Hospital for Active Treatment "Sveti Ivan Rilski", Sofia, Clinic of Clinical Hematology, Sofia
  - Multiprofile Hospital for Active Treatment - Sofia, part of Military Medical Academy, Clinic of Hematology, Sofia
  - Specialized Hospital for Active Treatment of Hematological Diseases, Sofia, Clinic of Hematology, Sofia
  - University Multiprofile Hospital for Active Treatment "Sveta Marina", Clinic of Clinical Hematology, Varna
- Canada (6):
  - University of Alberta Hospital, Edmonton, Alberta
  - Providence Hematology - Vancouver, Vancouver, British Columbia
  - Nova Scotia Health Authority, Centre for Clinical Research, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Research Institute, Odette Cancer Center, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Chile (5):
  - Dr. Guillermo Grant Benavente - Concepcion Regional Hospital, Concepción, Bio Bio
  - IC La Serena Research, La Serena, Coquimbo Region
  - SAGA Clinical Research Center SpA, Santiago
  - Clinic Inmunocel, Santiago
  - Center for Clinical Studies and Medical Research (CECIM), Santiago
- Czechia (4):
  - University Hospital Brno, Clinic of Internal Medicine - Hematology and Oncology, Brno
  - University Hospital Hradec Kralove, 4th Internal Clinic of Hematology, Hradec Králové
  - University Hospital Kralovske Vinohrady, Clinic of Internal Hematology, Prague
  - Institute of Hematology and Blood Transfusion, Division of Training and Development, Prague
- France (4):
  - Archet 1 and 2 hospital, Nice
  - Saint-Louis Hospital, Paris
  - Poitiers University Hospital Center - Miletrie Site, Poitiers
  - IUCT-Oncopole, Toulouse
- Germany (8):
  - University Hospital Bronn, Bonn, North Rhine-Westphalia
  - Marien Hospital Duesseldorf GmbH, Clinic for Oncology, Hematology and Palliative Medicine, Düsseldorf, North Rhine-Westphalia
  - University Hospital Leipzig, Clinic and Policlinic for Internal Medicine I Haematology and Stem Cell Therapy, Medical Oncology, Haemostaseology, Leipzig, Saxony
  - University Hospital Halle (Saale), Department of Internal Medicine IV - Hematology and Oncology, Halle, Saxony-Anhalt
  - University Clinic of Hematology, Oncology and Cell Therapy, Magdeburg, Saxony-Anhalt
  - UKSH, Lübeck, Schleswig-Holstein
  - Praxis am Volkspark Berlin, Berlin
  - Charite Universitatsmedizin Berlin, Berlin
- Hungary (5):
  - Semmelweis University, Department of Internal Medicine and Haematology, Division of Hematology, Budapest
  - University of Debrecen Clinical Center, Clinic of Internal Medicine, Department of Hematology, Debrecen
  - Mor Kaposi General Hospital, Department of Hematology, Kaposvár
  - Szabolcs-Szatmar-Bereg County Teaching Hospital, Department of Hematology, Nyíregyháza
  - Fejer County St. Gyorgy University Teaching Hospital, Department of Internal Medicine III, Hematology, Székesfehérvár
- India (13):
  - Heamto Oncology Clinic Ahmedabad Pvt. Ltd., Ahmedabad, Gujarat
  - Apollo Hospital International Ltd, Ahmedabad, Gujarat
  - Fortis Memorial Research Institute, Gurgaon, Haryana
  - Amrita Institute of Medical Sciences, Ernākulam, Kerala
  - Tata Memorial Centre, Mumbai, Maharashtra
  - Christian Medical College, Ludhianana, Ludhiana, Punjab
  - Christian Medical College, Vellore, Tamil Nadu
  - Max Super Speciality Hospital Vaishali (A Unit Of Crosslay Remedies Ltd.), Ghaziabad, Uttar Pradesh
  - NRS Medical College and Hospital, Kolkata, West Bengal
  - Tata Medical Center, Kolkata, Kolkata, West Bengal
  - Postgraduate Institute of Medical Education and Research, Chandigarh
  - Rajiv Gandhi Cancer Institute & Research Centre, Delhi
  - Medanta the Medicity, Gūrgaon
- Ireland (6):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Tallaght University Hospital, Dublin
  - St Vincent's University Hospital (SVUH), Dublin
  - University Hospital Limerick, Limerick
- Israel (4):
  - Hadassah Medical Center, Department of Hematology, Jerusalem
  - Rabin Medical Center, Davidoff Cancer Center, Hemato-Oncology Institute, Petah Tikva
  - Chaim Sheba Medical Center, Department of Hematology, Myelodysplastic Syndromes Center, Ramat Gan
  - The Tel Aviv Sourasky Medical Center, Department of Hematology and Bone Marrow Transplantation, Leukemia Service, Tel Aviv
- Italy (6):
  - Careggi University Hospital, Florence
  - Maggiore Polyclinic Hospital, Foundation IRCCS Ca' Granda, Milan
  - Polyclinic San Matteo, IRCCS, Department of Oncohematology, Operative Unit of Hematology, Pavia
  - Foundation PTV - Polyclinic Tor Vergata, Rome
  - Clinical Institute Humanitas, IRCCS, Rozzano
  - Institute of Cancer Research and Treatment of Candiolo, Turin
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Peru (5):
  - Edgardo Rebagliati Martins National Hospital, Lima, Jesus Maria
  - Anglo American Clinic, Lima, La Molina
  - IPOR: Peruvian Institute of Oncology & Radiotherapy, Lima, San Isidro Lima
  - Daniel Alcides Carrion National Hospital, Bellavista
  - National Institute of Neoplastic Diseases, Lima
- Poland (3):
  - Pratia Oncology Katowice, Katowice
  - Nicolaus Copernicus Provincial Multispecialty Oncology and Traumatology Center in Lodz, General Hematology Unit, Lodz
  - Clinical Hospital Of The Ministry Of Internal Affairs And Administration With Warmia And Mazury Oncology Centre In Olsztyn, Clinical Department of Hematology and Internal Medicine with Bone Marrow Transplantation Center, Olsztyn
- South Africa (4):
  - Haemalife, Cape Town
  - Capital Haematology Hospital, Durban
  - Charlotte Maxeke Johannesburg Academic Hospital, Hemophilia Comprehensive Care Center, Johannesburg
  - Alberts Cellular Therapy, Pretoria
- South Korea (6):
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Soon Chun Hyang University Hospital Seoul, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (6):
  - University Clinical Hospital of Salamanca, Department of Hematology, Salamanca, Castille and León
  - University Hospital Vall d'Hebron, Department of Hematology, Barcelona, Catalonia
  - Catalan Institute of Oncology, Hospital Duran i Reynals, Department of Clinical Hematology, L'Hospitalet de Llobregat, Girona
  - University Hospital Ramon y Cajal, Madrid, Madrid
  - University Hospital Foundation Jimenez Diaz, Madrid, Madrid
  - University and Polytechnic Hospital La Fe, Valencia, Valencia
- Sweden (2):
  - Karolinska University Hospital, Huddinge, Stockholm County
  - Skane University Hospital - Lund, Department of Hematology and Vascular Disorders, Lund
- Taiwan (6):
  - Changhua Christian Hospital, Changhua, Changhua County
  - Chang Bing Show Chwan Memorial Hospital, Changhua, Changhua County
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan
- Thailand (5):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Banphaeo General Hospital, Bangkok
  - Maharaj Nakorn Chiangmai Hospital, Chiang Mai
- Turkey (Türkiye) (7):
  - Adana City Hospital, Adana
  - Ankara Etlik City Hospital, Ankara
  - Ankara University Medical Faculty Cebeci Hospital, Ankara
  - Antalya Education and Training Hospital, Antalya
  - Mersin Medicalpark Hospital, Mersin
  - Sakarya University Medical Faculty Hospital, Sakarya
  - Ondokuz Mayis University School of Medicine, Department of Hematology, Samsun
- United Kingdom (8):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - St James's University Hospital, Leeds
  - King's College Hospital, London
  - Sarah Cannon Research Institute (SCRI), London
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.